CLINICAL TRIAL: NCT00254462
Title: Pharmacological Treatment of ADHD in Young Children
Brief Title: Atomoxetine for Treating Attention Deficit Hyperactivity Disorder in Young Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0164-03-FB; K23MH066127 (NIH)
Record Dates: First submitted 2005-11-14; First posted 2005-11-16 (Estimated); Results first posted 2013-07-17 (Estimated); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: ADHD; Atomoxetine
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- atomoxetine and parent training (Experimental): atomoxetine capsules, dose 0.5mg/kg/day to 1.8mg/kg/day administered once daily for 8 weeks
  Interventions: Drug: Atomoxetine; Behavioral: Parent Training
- placebo and parent training (Placebo Comparator): matching placebo capsules, dose 0.5mg/kg/day to 1.8mg/kg/day administered once daily for 8 weeks
  Interventions: Drug: Placebo; Behavioral: Parent Training

INTERVENTIONS:
Drug: Atomoxetine — Participants will receive atomoxetine for 8 weeks up to a maximum of 1.8 mg/kg/day. Dosed once daily in capsule formulation.
  Other Names: Strattera
  Arms: atomoxetine and parent training
Drug: Placebo — Participants will receive placebo for 8 weeks. Dosed once daily, capsule formulation.
  Other Names: Pill placebo
  Arms: placebo and parent training
Behavioral: Parent Training — All children will receive parent training for the duration of the study.
  Other Names: Psychosocial and educational intervention

SUMMARY:
This study will evaluate the effectiveness of atomoxetine in reducing the symptoms of attention deficit hyperactivity disorder (ADHD) in young children.

DETAILED DESCRIPTION:
Attention deficit hyperactivity disorder (ADHD) is one of the most common mental disorders in children. Children with ADHD often have impaired functioning in home and school and usually experience difficulty relating to peers. If left untreated, the disorder can have long-term adverse effects into adolescence and adulthood. Atomoxetine is a selective noradrenergic reuptake inhibitor that is FDA-approved for the treatment of ADHD in children, adolescents, and adults. Unlike most other medications for ADHD, atomoxetine is not a stimulant. Studies have shown that atomoxetine is effective in treating ADHD, but more information is needed on its effectiveness in young children. This study will evaluate the effectiveness of atomoxetine in reducing the symptoms of ADHD in young children.

Participants in this double-blind study will be randomly assigned to receive either atomoxetine or placebo for 8 weeks. In addition, all children will receive parent training for the duration of the study. For the first 5 weeks, participants will report to the study site weekly for assessments of ADHD symptoms. Study visits will occur every other week for the remainder of the study.

ELIGIBILITY:
Inclusion Criteria:

* Parent and child must be English speaking
* Child has been living with parent/guardian for at least six months
* Meets criteria for ADHD on the DISC, on clinical interview, and on clinical consensus conference
* ADHD is primary disorder with symptoms present for at least 9 months
* ADHD-IV-Rating Scale (ADHD-IV-RS)score that is at least 1.5 standard deviations above age and sex norms
* Score of 55 or below on the Children's Global Assessment Scale
* Score of 4 or greater on the Clinical Global Impression Scale
* Estimated Intelligence Quotient (IQ) of 70 or greater
* Currently participating in school at least 2 half-days per week
* Able to identify a teacher who can make valid assessments
* Patient and parent are able to attend regular study visits

Exclusion Criteria:

* Currently taking other psychotropic medications or other medications with effects on the central nervous system
* Currently being treated effectively with atomoxetine
* Major medical conditions that might interfere with study medications
* History of or current clinically significant kidney illness
* Evidence of adjustment disorder, autism, psychosis, bipolar disorder, suicide ideations, or any other psychiatric disorder requiring treatment with additional psychotropic medication
* History of physical, sexual, or emotional abuse impacting clinical presentation
* Prior failure to respond to an adequate trial of atomoxetine

Ages: 5 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 93 (Actual)
Dates: Start 2005-10-01 (Actual); Primary Completion 2008-08-01 (Actual); Study Completion 2008-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Kratochvil, MD, Principal Investigator — University of Nebraska
Locations (3):
- United States (3):
  - University of Nebraska Medical Center, Omaha, Nebraska
  - New York State Psychiatric Institute, New York, New York
  - Duke University Medical Center, Durham, North Carolina

REFERENCES:
- [Result] Kratochvil CJ, Vaughan BS, Stoner JA, Daughton JM, Lubberstedt BD, Murray DW, Chrisman AK, Faircloth MA, Itchon-Ramos NB, Kollins SH, Maayan LA, Greenhill LL, Kotler LA, Fried J, March JS. A double-blind, placebo-controlled study of atomoxetine in young children with ADHD. Pediatrics. 2011 Apr;127(4):e862-8. doi: 10.1542/peds.2010-0825. Epub 2011 Mar 21. PMID 21422081

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited in outpatient child psychiatry clinics at 3 academic institutions between October, 2005 and June 2008.
Pre-assignment Details: The ADHD diagnosis was confirmed using standardized measures and cases were reviewed on conference calls by professionals from all 3 sites.
Groups:
- Atomoxetine: Recommended dosing of once per day, with divided dosing allowed at investigators discretion. Maximum dose of 1.8 mg/kg/day.
- Placebo: Recommended dosing of once per day, with divided dosing allowed at investigators discretion.
Period: Overall Study
Arm/Group | Atomoxetine | Placebo
Started | 44 | 49
Completed | 36 | 39
Not Completed | 8 | 10

BASELINE CHARACTERISTICS:
Groups:
- Atomoxetine: Recommended dosing once daily, divided dosing at investigator discretion. Maximum dose of 1.8 mg/kg/day.
- Placebo: Recommended dosing once daily, divided dosing at investigator discretion.
- Total: Total of all reporting groups
Arm/Group | Atomoxetine | Placebo | Total
Number analyzed (Participants) | 44 | 49 | 93
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 44 | 49 | 93
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.1 (0.6) | 6.1 (0.5) | 6.1 (0.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 18 | 30
  Male | 32 | 31 | 63
Region of Enrollment [Number; unit: participants]
  United States | 44 | 49 | 93

OUTCOME MEASURES:

1. Primary Outcome: Change in ADHD-IV Rating Scale Total Score
Description: Measures 18 symptoms of attention deficit hyperactivity disorder (ADHD). Each symptom rated 0-3, for a minimum total score of 0, and a maximum total score of 54 for the scale. A higher score reflects more severe symptomatology.
  The inattentive subscale and the hyperactive/impulsive subscale each has a minimum score of 0 and maximum score of 27.
Time Frame: Measured at baseline and at Week 8. These are the only two timepoints calculated, later timepoint subtracted from earlier timepoint.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Atomoxetine: Recommended dosing once daily, allowed to give in divided dose at investigator discretion. Maximum dose of 1.8 mg/kg/day.
- Placebo: Recommended dosing once daily, allowed to give in divided dose at investigator discretion.
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 44 | 49
units on a scale | -13.2 (1.7) | -5.8 (1.2)

2. Secondary Outcome: Change in Total ADHD-IV Teacher
Description: Measures 18 symptoms of ADHD. Each symptom rated 0-3, for a maximum total score of 54 for the scale. A higher score reflects more severe symptomatology.
Time Frame: Measured at baseline and at Week 8. Later time point is subtracted from earlier time point.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Atomoxetine: Recommended dosing once daily, divided dose at investigator discretion. Maximum daily dose of 1.8 mg/kg/day.
- Placebo: Recommended dosing once daily, divided dose at investigator discretion.
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 44 | 49
units on a scale | -12.5 (1.7) | -5.0 (1.4)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Atomoxetine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/49
Other Adverse Events (participants affected / at risk) | 18/44 | 11/49
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atomoxetine (N=44) | Placebo (N=49)
aches/pains (General disorders) | 6 | 7
affective flattening/blunting (Psychiatric disorders) | 2 | 2
attention/hyperactivity (Psychiatric disorders) | 3 | 6
decreased appetite (Gastrointestinal disorders) | 13 | 4
dermatological (Skin and subcutaneous tissue disorders) | 6 | 5
disruptive behavior (Psychiatric disorders) | 3 | 4
gastrointestinal upset (Gastrointestinal disorders) | 17 | 8
insomnia (General disorders) | 1 (3) | 3 (10)
mood lability (Psychiatric disorders) | 18 (58) | 11 (22)
respiratory (Respiratory, thoracic and mediastinal disorders) | 5 | 4
sedation (General disorders) | 13 | 5
weight loss (General disorders) | 2 | 2

LIMITATIONS AND CAVEATS:
Study design does not allow differentiation between placebo response and psychoeducational treatment effect. Eight-week duration does not allow for examination of long-term effectiveness or assessment of adverse effects over time.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No